CLINICAL TRIAL: NCT06858917
Title: Comparison of Impar Ganglion Block and Sacral Erector Spinae Plane Block for Chronic Coccygodynia: a Randomized Controlled Trial
Brief Title: Comparison of Impar Ganglion Block and Sacral Erector Spinae Plane Block in Patients with Coccygodynia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Tuba Tanyel Saraçoğlu, Principal Investigator, Başakşehir Çam & Sakura City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22.05.2024.01
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-02

CONDITIONS: Coccygodynia; Coccydynia
Keywords: Coccygodynia; Coccydynia; impar block; sacral erector spinae plane block

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ganglion İmpar Block Group (Active Comparator): Participants in this group will performed ganglion impar block
  Interventions: Procedure: Ganglion Impar Block
- Sacral Erector Spinae Plane Block (Active Comparator): Participants in this group will performed sacral erector spinae plane block
  Interventions: Procedure: Sacral Erector Spinae Plane Block

INTERVENTIONS:
Procedure: Ganglion Impar Block — Block of the ganglion impar is performed by injecting a mixture of steroid and local anaesthetic in front of the sacrococcygeal joint. This procedure is performed in a sterile operating theatre under ultrasound and/or fluoroscopic (X-ray) guidance. Radiopaque agents are also used during the procedure to confirm the location.
  Other Names: impar block
  Arms: Ganglion İmpar Block Group
Procedure: Sacral Erector Spinae Plane Block — The sacral erector spina plan block is performed with ultrasound guidance by injecting a high volume mixture of local anaesthetic and steroid into the fascia under the erector spina muscles in the sacral region.
  Other Names: Sacral multifidus plane block
  Arms: Sacral Erector Spinae Plane Block

SUMMARY:
Coccygodynia is a condition that causes pain in the tailbone (coccyx) area. While it can develop after trauma, such as a fall or fracture, in some cases, no clear cause is identified. Patients who do not experience relief from standard treatments like pain medications, physical therapy, and posture adjustments may be referred to specialized pain management clinics for further treatment options.

Several interventional procedures can help manage coccygodynia. These include impar ganglion block, radiofrequency ablation, caudal epidural steroid injections, sacral erector spinae plane (ESP) block, and coccygeal nerve blocks. These procedures are commonly performed in pain treatment centers and aim to reduce discomfort by targeting specific nerves responsible for transmitting pain signals.

Impar ganglion block is one of the most frequently used treatments for coccygodynia. It involves injecting a local anesthetic, with or without steroids, into a small nerve cluster in front of the sacrococcygeal joint. This procedure is performed under ultrasound and/or fluoroscopic (X-ray) guidance in a sterile operating room setting to ensure accuracy and safety. While the goal is to relieve pain, potential risks include temporary worsening of pain, bleeding, infection, or, in rare cases, rectal injury.

Another interventional option is the sacral erector spinae plane (ESP) block, a technique that delivers local anesthetic under the erector spinae muscles in the sacrum. This procedure, also performed under ultrasound guidance in a sterile environment, is used to block pain signals from the coccyx and surrounding areas. Like the impar ganglion block, it can be effective for pain relief, but possible side effects include temporary pain increase, bleeding, and infection at the injection site.

Both procedures are minimally invasive.

DETAILED DESCRIPTION:
Coccygodynia is defined as pain localized in the coccygeal region. While previous trauma and fractures may contribute to its development, in many cases, no identifiable etiology can be determined. Patients who continue to experience pain despite conservative treatment and physiotherapy are often referred to pain management outpatient clinics for interventional treatment options. Various interventional procedures are utilized in the management of coccygodynia, including impar ganglion block and radiofrequency applications, caudal epidural steroid injections, sacral erector spinae plane block, and coccygeal nerve blocks, all of which are commonly performed in pain treatment clinics. Impar ganglion block is administered under sterile conditions in the sacrococcygeal region within an operating room setting, utilizing ultrasound and/or fluoroscopic guidance. This procedure aims to alleviate pain; however, potential complications include increased pain, bleeding at the procedural site, rectal perforation, and infection. Sacral erector spinae plane block is another interventional approach performed under sterile conditions in the operating room using ultrasound guidance. Similar to the impar ganglion block, its primary objective is pain reduction, though it also carries risks such as increased pain, bleeding, and infection at the procedural site

ELIGIBILITY:
Inclusion Criteria:

* Those who have had chronic coccygodynia for at least 3 months
* Being between the ages of 18-65
* Patients who do not respond to conservative treatments (analgesics, physical therapy modalities etc.) and are scheduled for interventional pain procedures

Exclusion Criteria:

* Patients who have undergone surgery to the coccyx region
* Having undergone an interventional pain procedure in the lumbar, sacral and coccyx regions within the last year
* Patients with systemic infection, local infection at the application site, and coagulopathy
* Pregnant and breastfeeding patients
* Having endocrine or rheumatological disease that may affect the musculoskeletal system in the relevant region and lead to diagnostic complexity (such as spondyloarthropathy)
* Patients with musculoskeletal system pathology that may contribute to symptoms in the relevant region and affect the evaluation of treatment results (such as lumbar disc herniation, sacroiliitis, spinal stenosis)
* Those with lumbar, sacral or coccygeal vertebra fractures
* Those with a history of allergic reactions to the contents of the injectate to be administered during an interventional pain procedure (especially contrast agent and local anesthetic)
* Those with mental disorders that may affect the evaluation during the follow-up periods during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale | Preprocedural, Week 1, Week 4, Week 12
  The Numeric Rating Scale (NRS) is an 11-point scale (0-10) used to assess pain intensity, with 0 indicating 'no pain' and 10 representing 'worst possible pain.

SECONDARY OUTCOMES:
Short Form-12 | Preprocedural, Week 1, Week 4, Week 12
  The Short Form-12 (SF-12) is a validated questionnaire assessing health-related quality of life. It generates separate Physical Component Summary (PCS) and Mental Component Summary (MCS) scores, where higher scores indicate better physical and mental health, while lower scores reflect poorer health status.
Pain-free sitting duration | Preprocedural, Week 1, Week 4, Week 12
  Patients will be asked to assess and record their pain-free sitting durations on the hard and soft surfaces they regularly use during pre-procedural and post-procedural follow-ups. They will be specifically instructed to perform these assessments using the same hard and soft surfaces each time.
Oswetry Disability Index | Preprocedural, Week 1, Week 4, Week 12
  The Oswestry Disability Index (ODI) was used to assess the degree of disability. The ODI consists of 10 items, evaluating pain intensity, personal care, lifting, walking, sitting, standing, social life, sleeping, traveling, and pain-related distress.

CONTACTS AND LOCATIONS:
Overall Officials: Tuba Tanyel Saraçoğlu, Principal Investigator — Başakşehir Çam & Sakura City Hospital
Locations (1):
- Başakşehir Çam and Sakura City Hospital, Istanbul, Başakşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No